CLINICAL TRIAL: NCT03571698
Title: Istanbul University, Faculty of Health Science, Division of Physiotherapy and Rehabilitation
Brief Title: The Efficacy of Exercise and Alternative Applications of NMES on Pain and Function in Patients With Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ekin Aktay, Physical Therapist Master in Science, Istanbul University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IstU
Record Dates: First submitted 2018-05-30; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Neuromuscular Electrical Stimulation; Exercise; Pain; Function
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise programme only (No Intervention): The treatment group received only exercise programme. The exercises was done by a physical therapist in clinical center. The treatment group received exercise programme with simultaneously active contraction with NMES with large electrodes.
- Exercise with NMES standard electrodes (Active Comparator): The treatment group received exercise programme with simultaneously active contraction with NMES with standard electrodes.The exercises was done by a physical therapist in clinical center. The treatment group received exercise programme with simultaneously active contraction with NMES with large electrodes.
  Interventions: Device: Neuromuscular Electrical Stimulator
- Exercise with NMES large electrodes (Active Comparator): The treatment group received exercise programme with simultaneously active contraction with NMES with large electrodes.The exercises was done by a physical therapist in clinical center. The treatment group received exercise programme with simultaneously active contraction with NMES with large electrodes.
  Interventions: Device: Neuromuscular Electrical Stimulator

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulator — The treatment group received exercise programme with simultaneously active contraction with NMES with large or standart electrodes.
  Arms: Exercise with NMES large electrodes; Exercise with NMES standard electrodes

SUMMARY:
The aim of the study was to investigate the efficacy of exercise and different size electrodes of neuromuscular electrical stimulation (NMES) applications on pain, range of motion (ROM), muscle strength, function status and depression in knee osteoarthritis.

60 voluntary patients were included in the study and these patients divided into three groups randomly. For Group 1 only exercise, for Group 2 simultaneously active contraction with NMES with standard size electrodes, for Group 3 simultaneously active contraction with NMES with large electrodes applied for 3 days per week, 18 session. Pain was measured with Visual analog Scale (VAS), ROM was measured with digital goniometer, muscle strength was measured with "Hand-held" dynamometer (Lafayette Instrument®, Lafayette, IN), functional status were measured with WOMAC (Western Ontario and McMaster Universities) Index and stair climbing test, balance was analysed with one leg standing test, depression was scored with Hospital Anxiety Depression Scale and patients satisfaction was scored with Global Rating Change Scales. The cases evaluated before and after treatment.

DETAILED DESCRIPTION:
Aim: This study investigated the effect of neuromuscular electrical stimulation (NMES) was applied with different size electrodes on the functionality, pain, range of motion (ROM), and muscle strength in patients wtih knee osteoarthritis (OA).

Material and Metod: Sixty patients with knee OA who received physical therapy for knee pain and functional disability at Istanbul University, Faculty of Health Sciences, Division of Physiotherapy were included. These patients divided into three groups randomly. Group 1 applied exercise programme. Group 2 performed exercise programme with NMES with standard size electrodes (5×5 cm²). Group 3 performed exercise programme with NMES with large size electrodes (10×20 cm², 3×18 cm², 10 3×7.5 cm², 7×14 cm²) NMES was applied for 20 minutes to Group 2 and Group 3. The patients attended 18 treatment sessions 3 times per week in the physical therapy clinic and underwent assesment before treatment and after 6 weeks of treatment. Pain was measured with Visual Analog Scale (VAS), range of motion (ROM) was measured with digital goniometer, muscle strength was measured with ''Hand-held'' dynomometer, functional status were measured with WOMAC (Western Ontario and McMaster Universities) Index and stair climbing test, balance was analysed with one leg standing test. Patients satisfaction was scored with Global Change Scales.

ELIGIBILITY:
Inclusion Criteria:

Acceppting to participate Being between 45-74 years according to the description of the World Health Organisation Being women Having Osteoarthritis on right knee. Having the symptoms of Grade 2-3 according to Kellgren ve Lawrence Classification Having a value below 30 according to Body Mass Index

Exclusion Criteria:

Not accepting to partipate Having left knee Osteoarthritis Having an orthopedic problem on lower extremity Having uncontrollable hypertension Having arteriovenous problem on lower extremity Having confusion about regular participation Having a neurogical problem Having learning and perception problem Having heart implant Being included in physiotherapy and rehabilitation program for knee OA in last 6 month Having injection application for knee in last 6 month

Ages: 47 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Visual Analoque Scale | The rest, night time and pain in activity were assessed by VAS before treatment versus after 6 weeks of treatment.
  Pain intensity was assessed using the VAS; each patient was asked the pain during the rest, activity, and at night time.
Knee Extensor Muscle Strength | Quadriceps Femoris Muscle strength was measured before treatment versus after 6 weeks of treatment.
  Quadriceps Femoris Muscle strength was measured using a Hand-held Dynomometer.

SECONDARY OUTCOMES:
Knee Range of Motion | Knee Flexion and extension were measured with Digital Goniometer on sitting position before treatment versus after 6 weeks.
  Knee Flexion and extension were measured using a Digital Goniometer.
Knee Range of Motion | Knee Flexion and extension were taken using Digital Goniometer before treatment versus after 6 weeks treatent.
  Knee Flexion and extension were taken using a Digital Goniometer on sitting position.
Muscle Strength using a Hand-held Dynomometer | Hip flexor, extensor, adductor, abductor groups muscles, knee flexor groups muscles strength were measaured before treatment versus after 6 weeks of treatment.
  Hip flexor, extensor, adductor, abductor groups muscles, knee flexor groups muscles strength were measaured using a Hand-held Dynomometer.
WOMAC (Western Ontario and McMaster Universities Index) | Pain, stiffness and physical function were assessed by WOMAC before treatment versus after 6 weeks of treatment.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:[1]
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.
Stair Climbimg Test (SCT) | Balance was assessed by SCT before treatment versus after 6 weeks of treatment.
  The SCT assesses the ability to ascend and descend a flight of stairs, as well as lower extremity balance.Test included the number of steps, the task requirement (ascent only or ascent/decent combined), or whether the test is timed over a set number of steps or the step count is recorded for a set period of time: 9-step ascend/descend, 4-step ascend/descend (6),3-step ascent cycle duration, 30-second test (12 steps), 3-step measured on 0 - 6 scale of level of assistance., and 6-step fast and self-paced.
One Leg Standing Test | Balance was assessed by One Leg Standing Test before treatment versus after 6 weeks of treatment.
  One single-leg standing was assessed balance. Test required the subject to stand with arms by his/her side.Timing was started when the subject raised one foot off the ground. Timing was stopped if the subject displaced the weight-bearing foot, touched the suspended foot to the ground, used the suspended limb to support the weight-bearing limb, or reached the maximum balance time of 30 seconds.
Global Rating Change Scales | Satisfactions was assessed using by Global Rating Change Scales before treatment versus after 6 weeks of treatment.
  Rating levels of satisfaction is critical to a successful survey. Global Rating Scale's levels of satisfaction may vary from "Not at all satisfied" to "Very Satisfied" or "Extremely Satisfied," but the scale is not balanced in the same way as Performance or Expectation.

CONTACTS AND LOCATIONS:
Overall Officials: Yıldız Analay Akbaba, Assist Prof., Study Director — Istanbul University; Ekin Aktay, MSc, Principal Investigator — Istanbul University

IPD SHARING:
Plan to Share IPD: No